CLINICAL TRIAL: NCT03421626
Title: Clinical Evaluation of the Xpert BCR-ABL Ultra Assay on the GeneXpert Instrument Systems
Brief Title: Clinical Evaluation of a Test for Monitoring Patients Diagnosed With Chronic Myeloid Leukemia (CML)
Status: Completed | Type: Observational
Sponsor: Cepheid (Industry)
Responsible Party: Sponsor
Other Study IDs: 231
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2018-01

CONDITIONS: Leukemia, Myelogenous, Chronic
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Primary Enrollment: Initial enrollment of patients with history of CML
  Interventions: Device: Xpert BCR-ABL Ultra

INTERVENTIONS:
Device: Xpert BCR-ABL Ultra — Semi-quantitation of BCR-ABL transcript in patients that have been previously diagnosed with CML

SUMMARY:
The objective of this study is to establish the performance of an assay that detects mRNA transcript levels in patients diagnosed with CML. The study is conducted at locations within the United States. Testing is performed on peripheral blood specimens provided by eligible enrolled patients. Results from this study will not be used for patient management decisions.

ELIGIBILITY:
Inclusion Criteria:

* prospective specimens:

  * Patient is at least 18 years of age
  * Patient has provided documented informed consent as required by the reviewing IRB. Experimental Bill of Rights will also be documented for all subjects enrolled in applicable states.
  * Patient has been diagnosed with CML.
  * Patient consents to provide at least 12 mL of peripheral blood for study purposes
* frozen specimens:

  * Specimen is from a subject diagnosed with CML
  * Specimen meets the manufacturer's criteria to support testing by both diagnostic assays

Exclusion Criteria:

* prospective specimens:

  * Patient is considered to be of insufficient health to supply the required volume of peripheral blood by his/her health care provider
  * Patient has been previously enrolled
* frozen specimens: • Specimen previously enrolled

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females at least 18 years of age who were previously diagnosed with CML from primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Method comparison to an on-market molecular diagnostic assay | Baseline = testing upon enrollment
  Comparison of Xpert to an on-market test for the quantitation of BCR-ABL

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - St. Alphonsus Regional Medical Center, Boise, Idaho
  - WJB Dorn VA Medical Center, Columbia, South Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Marshfield Clinic, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No